CLINICAL TRIAL: NCT00448162
Title: The Chinese Mutation Hotspot of ENaC Causing Liddle's Syndrome and the Association of ENaC Variations and Hypertension
Status: Suspended | Type: Observational
Why Stopped: no enough fund
Sponsor: Peking Union Medical College (Other)
Responsible Party: Rutai Hui, Fuwai Hospital
Other Study IDs: SGL-032-01
Record Dates: First submitted 2007-03-15; First posted 2007-03-16 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2009-05

CONDITIONS: Hypertension
Keywords: hypertension, ENaC, Liddle's syndrome, variation
MeSH Terms: conditions — Hypertension; Liddle Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The variations of ENaC have an impact on the degradation of epithelial sodium channels and sodium reabsorption, and thus are associated with hypertension and hypokalemia.

Liddle's syndrome is a rare monogenic form of autosomal-dominant hypertension caused by truncating or missense mutations in the C-termini of epithelial sodium channel β- or γ-subunit encoded by SCNN1B or SCNN1G. Our purpose is to determine the hotspot of mutation causing Chinese Liddle's syndrome.

The second purpose is to determine wether the polymorphisms of ENaC are associated with hypertension in Chinese. Some polymorphisms of ENaC associated with hypertension may be genetic risk factors for Chinese hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypertension and Liddle's syndrome
* Clinical diagnosis of normal controls with no cardiovascular disease

Exclusion Criteria:

* Hypertension caused by other single gene mutation

Ages: 8 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients were defined as being hypertensive if they had systolic and/or diastolic BP levels >=140/90mm Hg on three occasions within 2 months and if they were without any antihypertensive treatment, and/or if they had been diagnosed as being hypertensive in the past and were currently receiving antihypertensive medications. The normotensive controls were defined as having systolic and/or diastolic BP levels <130/85mm Hg and with no family history of hypertension. Patients were excluded when they had any known renal diseases or secondary hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2005-05; Study Completion 2009-12

CONTACTS AND LOCATIONS:
Overall Officials: Rutai Hui, PhD, MD, Study Director — Key Laboratory for Clinical Cardiovascular Genetics, Ministry of Education, China & Sino-German Laboratory for Molecular Medicine,
Locations (1):
- FuWai Hospital, Beijing, Beijing Municipality, China